CLINICAL TRIAL: NCT05632497
Title: Study of Translational Process of Relationship Between Intestinal Microbiota of Dysbiosis and the Psychic Symptoms of Anorexia Nervosa (Eating Disorders and Anxio-depression Disorders)
Brief Title: Alteration of Symbiosis Intestinal Microbiota on Patients With Anorexia Nervosa
Acronym: INT-METAVOSA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211375; 2021-A02529-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-11-14; First posted 2022-11-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa; Dysbiosis; Anxious Depression
Keywords: Anorexia nervosa; Dysbiosis; Anxious depression; Intestinal microbiota; Body mass index
MeSH Terms: conditions — Anorexia Nervosa; Dysbiosis | interventions — Defecation; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample will be collected for all of 2 types of subjects (patients and health volunteers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia patients: Hospitalized anorexia patients with body mass index < 15.
  Interventions: Biological: Stool and blood samples
- Healthy controls: Health volunteers: 18 years or older with body mass index between 18.5 and 25.
  Interventions: Biological: Stool and blood samples

INTERVENTIONS:
Biological: Stool and blood samples — Stool and blood samples

SUMMARY:
The purpose of this study will be to study the association between the level of psychic symptomatic of anorexia nervosa (AN) (intensity of food restriction, symptoms of anxiety and depression) and alteration of host environment symbiosis and the mechanism (dysbiosis of intestinal microbiota, increase of intestinal permeability, immunity alteration and low-grade inflammation).

DETAILED DESCRIPTION:
This is a monocentric study aims to characterise the intestinal microbiota of anorexia nervosa patients with malnutrition, in comparison with the control subject, by DNA sequencing and metagenomic method. The interaction of intetinal microbiota with the host will be studied through the mecanistic studies and various parameters of alteration of symbiosis (intestinal permeability, inflammation) and their association with psychic symptoms of anorexia nervosa.

The objective of this approche is to have not only a descrition of genomic of material of sampling, but also an overview of its potential functioning.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patients aged ≥18 years;
* Anorexia according to DSM-5 and CIDI (Composite International Diagnostic Interview);
* Body mass index (BMI) (P/T2) < 15;
* Hospitalization for nutrition rehabilitation;
* Covered by a health insurance;
* Informed consent form signed.

For Healthy Volunteers:

* Aged ≥18 years;
* 18.5 < BMI (P/T2) < 25;
* Covered by a health insurance;
* Informed consent form signed.

Exclusion Criteria:

For patients:

* Patients no-responding all criteria of DSM-5 or CIDI scores;
* Taken of antibiotic treatment 2 months / or laxativ 3 weeks before hospitalization;
* Somatic comorbidity should perturb intestinal microbiota (Crohn's disease, diabetes and all other chronic inflammatory diseases);
* Patients under guardianship;
* Patients covered by french AME scheme.

For Healthy Volunteers:

* Any disease should perturb intestinal microbiota;
* Recent ponderal variation;
* Taken of antibiotic treatment 2 months or laxativ 3 weeks before hospitalization;
* Under guardianship;
* Covered by french AME scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with anorexia nervosa for nutrition rehabilitation in the department of nutrition in Paul Brousse hospital (Villejuif) - APHP.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder | at baseline
  By Eating Disorder Inventory (EDI-3)
Anxio-depressive symptomatologic assessements by HAD score | at baseline
  By HAD score
Anxio-depressive symptomatologic assessements by scale of Beck BDI 13 | at baseline
  By scale of Beck BDI 13
Anxio-depressive symptomatologic assessements by LSAS Lieboweitz social anxiety scale | at baseline
  By LSAS Lieboweitz social anxiety scale
Anxio-depressive symptomatologic assessements by MOCI | at baseline
  By Maudsley Obsessions and compulsions inventory (MOCI).
Anxio-depressive symptomatologic assessements | at baseline
  By HAD score, scale of Beck BDI 13, LSAS Lieboweitz social anxiety scale, Maudsley Obsessions and compulsions inventory (MOCI).
Physical exercise | at baseline
  By Global physical activity questionnaire (GPAQ)
Biological parameter | at baseline
  By serum serotonin level

SECONDARY OUTCOMES:
Diversity indice | at baseline
  By index de Sympson et Shannon
Intestinal permeability | at baseline
  By serum zonulin level
Immunity alteration | at baseline
  By interleukins and CRP level
Liver function | at baseline
  Cytolyse analysis in serum
BMI | at baseline
  Calculate of BMI.
Body composition | at baseline
  By Dexa-Scan.
Energy expenditure | at baseline
  Calculate of indirect calorimetry and blood parameters
Intestinal functional disorders | at baseline
  By Francis scale, ,transit with pellets and abdomen x-ray
Gene and species richness | at baseline
  By 16S rRNA gene sequencing method and Metagenomics
Circulating mitochondrial DNA copy number | at baseline
  By telemore size and HLA genotyping
Heart damage | at baseline
  By Left Ventricle Ejection Fraction < 50% structural parameters on ultrasound
Presence of Autistic symptoms (1) | at baseline
  By Glasgow Sensory Questionnaire GSQ)
Presence of Autistic symptoms (2) | at baseline
  By The SWedish Eating Assessment for Autism spectrum disorders GSQ)
EDI | at baseline
  QUESTIONNAIRE EDI or EATING DISORDER INVENTORY (Eating disorder inventory 2nd edition (EDI-2)
Eating Disorder Diagnostic | at baseline
  By Eating Disorder Diagnostic Scale (EDDS)-DSM-5 VERSION (2015 Wiley Periodicals)
Eating behaviors assessment | at baseline
  By the Detail and Flexibility Questionnaire (DFlex).

CONTACTS AND LOCATIONS:
Overall Officials: Mouna HANACHI GUIDOUM, MD, Principal Investigator — Service de Nutrition Clinique, Hôpital Paul Brousse - APHP
Locations (1):
- Service de Nutrition Clinique, Hôpital Paul Brousse (APHP), Villejuif, France